CLINICAL TRIAL: NCT00145132
Title: Serotonin and Dopamine Transporter (SERT, DAT) Availabilities as Assessed by b-CIT and SPECT, and Neurophysiological Measures of Central Serotonergic Activity in Patients With Depression Under Treatment With Escitalopram
Brief Title: Beta-CIT-SPECT and Neurophysiology in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Oliver Pogarell, MD, University of Munich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ESCIT-SPECT-Pogarell; EK287/98
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Depression
Keywords: depression; β-CIT-SPECT; SERT; DAT; neurophysiology; LDAEP; escitalopram; SSRI
MeSH Terms: conditions — Depression

INTERVENTIONS:
Procedure: β-CIT-SPECT, Neurophysiology — β-CIT-SPECT scans and EEG recordings, two assessments each

SUMMARY:
Aim of this project is to investigate the effects of escitalopram on monoamine transporter (SERT, DAT) availabilities as assessed by b-CIT and SPECT, and on neurophysiological parameters such as the loudness dependence of auditory evoked potentials (LDAEP) in patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric in or outpatients with acute depressive episode
* Indication for pharmacological treatment

Exclusion Criteria:

* Acute suicidality
* Neurological or severe somatic disorders
* Occupational exposition to radiation >15 mSv per year
* Women during pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
changes in β-CIT/neurophysiological measurements from baseline to week 4 | two assessments, at baseline and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Pogarell, MD, Principal Investigator — Dept. of Psychiatry, University of Munich
Locations (1):
- Depts. of Psychiatry and Nuclear Medicine, Ludwig-Maximilians-University of Munich, Munich, Germany